CLINICAL TRIAL: NCT02754986
Title: Quantification of Autonomic Nervous Activity by Heart Rate Variability and Approximate Entropy in High Ultrafiltration Rate During Hemodialysis
Brief Title: Quantification of Autonomic Nervous Activity During Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hyogo (Other)
Responsible Party: Principal Investigator, Yoshihiro Tsuji, clinical engineer, University of Hyogo
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UHyogo
Record Dates: First submitted 2016-03-01; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Kidney Disease on Hemodialysis
Keywords: heart rate variability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- measuring Holter electrocardiogram (Experimental): Hotter ECG will be recorded continuously during hemodialysis
  Interventions: Other: Analysis of the holter electrocardiogram

INTERVENTIONS:
Other: Analysis of the holter electrocardiogram
  Other Names: Analysis of heart rate variability with using holter electrocardiogram

SUMMARY:
This study assesses autonomic nervous system function by power spectral analysis of RR interval dynamics in ultrafiltration subjects without blood pressure variation.

DETAILED DESCRIPTION:
Variations over time in autonomic nervous activity due to differences in ultrafiltration rate will be evaluated by measuring heart rate variability in hemodialysis patients without blood pressure variations during HD session.

The subjects will be divided into 3 groups, those with UFR < 10 ml/hr/kg; ≥10 ml/hr/kg but ≤ 15 ml/hr/kg; and >15 ml/hr/kg, and Holter ECG are recorded continuously during HD session using frequency analysis of RR intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable undergoing hemodialysis without hanging in blood pressure during hemodialysis.

Exclusion Criteria:

* Patients with chronic atrial fibrillation
* Patients with frequent ventricular premature beats
* Patients with a permanent pacemaker
* Patients with taking antihypertensive drugs
* Patients with medical treatment due to changes in blood pressure

Max Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The outcome measures was low frequency power (LF, ms2) to high frequency power (HF, ms2) ratio (LF/HF ratio) of heart rate variability. The three subject groups with difference ultrafiltration were compared by LF/HF ratio during hemodialysis session. | 4 hours
  Variations over time in autonomic nervous activity due to differences in ultrafiltration rate will be evaluated by measuring heart rate variability.

CONTACTS AND LOCATIONS:
Overall Officials: Yuko Mizuno-Matsumoto, Ph.D., Study Director — Graduate School of Applied Informatics, University of Hyogo
Locations (1):
- Graduate School of Applied Informatics, University of Hyogo, Kobe, Hyōgo, Japan

IPD SHARING:
Plan to Share IPD: Yes